CLINICAL TRIAL: NCT06794684
Title: Evaluation of Atherosclerotic Plaque Progression by Coronary Computed Tomography Angiography and Intracoronary Imaging Techniques in Patients With Coronary Artery Disease
Brief Title: PRogression of Atheroma Evaluated by CT Angiography and IntraCoronary Imaging tEchniques
Acronym: PRACTICE
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, Professor, Ruijin Hospital
Other Study IDs: RJH-PRACTICE
Record Dates: First submitted 2025-01-14; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Coronary Arterial Disease (CAD); Coronary Arteriosclerosis
Keywords: Coronary CTA; Plaque Progression; coronary artery disease; high-risk plaques; plaque composition; intracoronary imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood sample at baseline and follow-up
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PRACTICE cohort: Subjects with CAD detected by coronary CTA are consecutively enrolled. All the patients will undergo clinical follow-up for up to 5 years. Repeat coronary CTA will be conducted after 2 years.

SUMMARY:
This is a combined cohort study with retrospectively and prospectively enrolled coronary artery disease (CAD) patients. All the patients will undergo clinical follow-up for up to 5 years, and repeat coronary CTA will be conducted after 2 years. Comprehensive morphological and functional plaque analysis will be performed. The impact of these morphological and functional parameters, alongside cardiometabolic factors and pharmacological treatments on plaque progression and the occurrence of major adverse cardiovascular events (MACEs) will be analyzed. In addition, intracoronary imaging techniques will be used to improve the accuracy of plaque analysis by coronary CTA.

DETAILED DESCRIPTION:
This is a combined cohort study with retrospectively and prospectively enrolled patients. Subjects with CAD detected by coronary CTA are consecutively enrolled. All the patients will undergo clinical follow-up for up to 5 years. Repeat coronary CTA will be conducted after 2 years. For patients referred to invasive coronary angiography, intracoronary imaging techniques, such as intravascular ultrasound (IVUS), optical coherence tomography (OCT), and near infrared spectroscopy (NIRS) will be performed. For all the prospectively enrolled patients, plasma and serum blood samples will be collected.

The purpose of this study is to investigate the natural history of coronary atherosclerotic plaques in this population. Comprehensive morphological plaque analysis will be performed to evaluate total atheroma volume (TAV), percent atheroma volume (PAV), plaque composition, high risk plaque features, and characteristics of perivascular adipose tissue (PVAT). Functional analysis will also be conducted to calculate hemodynamic parameters such as wall shear stress (WSS), oscillatory shear index (OSI), relative residence time (RTT), transverse WSS (transWSS), axis plaque stress (APS), fractional flow reserve (FFR), and δFFR across lesions. The associations of these morphological and functional parameters with plaque progression and the onset of major adverse cardiovascular events (MACEs) will be analyzed. In addition, the impact of pharmacological treatments and the levels of cardiometabolic factors on coronary plaque progression will also be investigated.

In the subpopulation who also receive intracoronary imaging examinations, intracoronary imaging modalities will be used to refine the inner and outer vessel contours, improve the accuracy of plaque composition characterization, and aid in the discovery of novel high-risk plaque features by coronary CTA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinically significant angina pectoris, or suspected CAD
* Receive coronary CTA scan, with a visible plaque (defined as ≥25% diameter stenosis) in major coronary arteries.

Exclusion Criteria:

* Unsuitable for coronary CTA (such as severe renal impairment, uncontrolled thyroid condition, allergic to iodine, etc.)
* Receive percutaneous coronary intervention (PCI) within 6 months
* Prior history of myocardial infarction or heart failure
* Prior history of percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
* Abnormal liver function (serum alanine aminotransferase [ALT] level exceeding 3 times the upper limit of normal) or abnormal kidney function (eGFR ≤30 ml/min)
* Familial hypercholesterolemia
* Estimated survival ≤ 1 year
* Malignant tumor
* Pregnant or lactation, or have the intention to give birth within one year
* Poor coordinance, unable to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a combination of retrospective and prospective cohort studies. Patients with clinical angina pectoris or suspected CAD who undergo coronary CTA scan, including outpatient and hospitalized patients, are consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in total atheroma volume (TAV) | 24 months
  changes in TAV in whole heart and in target lesions measured by coronary CTA and quantification analysis at baseline and during follow-up

SECONDARY OUTCOMES:
Major cardiovascular events (MACEs) | 5 years
  A composite endpoint of cardiovascular death, non-fatal myocardial infarction, and unplanned revascularization during follow-up
Cardiovascular death | 5 years
  The occurrence of cardiovascular death during follow-up
Myocardial infarction | 5 years
  The occurrence of myocardial infarction during follow-up
Unplanned revascularization | 5 years
  The occurrence of unplanned revascularization during follow-up
Changes in calcified plaque volume | 24 months
  Changes in calcified plaque volume in whole heart and in target lesions measured by coronary CTA and quantification analysis at baseline and during follow-up
Changes in non-calcified plaque volume | 24 months
  Changes in non-calcified plaque volume in whole heart and in target lesions measured by coronary CTA and quantification analysis at baseline and during follow-up
Changes in fibrous plaque volume | 24 months
  Changes in fibrous plaque volume in whole heart and in target lesions measured by coronary CTA and quantification analysis at baseline and during follow-up
Changes in fibrousfatty plaque volume | 24 months
  Changes in fibrousfatty plaque volume in whole heart and in target lesions measured by coronary CTA and quantification analysis at baseline and during follow-up
Changes in necrotic core volume | 24 months
  Changes in plaque necrotic core volume in whole heart and in target lesions measured by coronary CTA and quantification analysis at baseline and during follow-up
Changes in high-risk plaque (HRP) features | 24 months
  Changes in the number of HRP features in whole heart and in target lesions measured by coronary CTA at baseline and during follow-up.
Changes in perivascular adipose tissue (PVAT) volume | 24 months
  Changes in the volume of PVAT measured by coronary CTA and quantification analysis at baseline and during follow-up
Changes in perivascular adipose tissue (PVAT) density | 24 months
  Changes in the density of PVAT measured by coronary CTA and quantification analysis at baseline and during follow-up
Changes in perivascular adipose tissue (PVAT) distribution | 24 months
  Changes in the distribution of PVAT measured by coronary CTA and quantification analysis at baseline and during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ruiyan Zhang, M.D., Ph.D., Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - CAAC East China Aviation Personnel Medical Appraisal Center, Civil Aviation Shanghai Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided